CLINICAL TRIAL: NCT04378803
Title: Mindfulness Training for Older Adults During the COVID-19 Pandemic
Brief Title: Mindfulness Training for Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ekaterina Denkova, Research Assistant Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 20200443
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Well Aging

STUDY DESIGN:
Intervention Model Description: The wait-list control group will receive the training program at a later point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness training (MT) group (Experimental): Receives 4 weeks of mindfulness training followed by a testing session. Then, 4 weeks of no-training interval followed by a testing session.
  Interventions: Behavioral: Mindfulness training (MT) Connect
- Wait-list control (WLC) group (Experimental): Receives 4 weeks of no-training interval followed by a testing session. Then, 4 weeks of mindfulness training followed by a testing session.
  Interventions: Behavioral: Mindfulness training (MT) Connect

INTERVENTIONS:
Behavioral: Mindfulness training (MT) Connect — MT Connect will involve instructor-led weekly sessions and mindfulness exercises over a 4-week interval for a total of 8 to 10 hours. There will be one instructor-led session per week that will last between 2 and 2.5 hours. Participants will also be asked to complete three categories of mindfulness exercises (formal and informal mindfulness exercises, and reflective practices) as part of their daily 'out-of-class' homework. The daily homework will require between 10 to 30 minutes to complete.

SUMMARY:
The purpose of this research study is to learn more about how mindfulness training may influence thinking and feeling.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are between 60 and 95 years of age
* Individuals who are fluent English speakers
* Individuals who are able to adequately and independently use electronic devices, such as a laptop, computer, or tablet, and have an Internet connection
* Individuals who are willing and able to consent to participate in the study

Exclusion Criteria:

* Individuals who are cognitively impaired and not independent in daily activities, such as the use of the telephone, preparing meals
* Individuals with an active and untreated mental condition (e.g., Bipolar disorder, Major Depression) and/or hospitalization for psychological/mental health issues within the last month.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Change in mindfulness skills as measured by Five-Facet Mindfulness Questionnaire (5FMQ) | Baseline to week 10
  5FMQ is a 15-item questionnaire with 5 sub-scales: observing, describing, acting with awareness, non-judgmental inner experience, and non-reactivity. The score for each sub-scale ranges from 3 to 15, a higher score is indicative of greater mindfulness skills.
Change in mindfulness skills as measured by decentering - Experiences Questionnaire (EQ). | Baseline to week 10
  EQ Decentering is an 11-item sub-scale measuring various thoughts and experiences, and the tendency to distance from those. The decentering score ranges from 1 to 55, with a higher score indicating high level of decentering.
Change in psychological health as measured by Patient Health Questionnaire 4 items (PHQ4). | Baseline to week 10
  PHQ4 is an ultra-brief 4-item measure of depression and anxiety with the total score ranging from 0 to 12. Higher score indicates higher level of anxiety and depression.
Change in positive affect on psychological health as measured by the short variant of the Positive and Negative Affect Scale (PANAS). | Baseline to week 10
  The PANAS positive sub-scale includes 5 items with a score ranges from 5 to 25 with a higher score indicating a higher positive mood.
Change in negative affect on psychological health as measured by the short variant of the Positive and Negative Affect Scale (PANAS). | Baseline to week 10
  The PANAS negative sub-scale includes 5 items with a score ranges from 5 to 25 with a higher score indicating a higher negative mood.
Change in loneliness measured by the loneliness questions from the social isolation battery. | Baseline to week 10
  The 3 loneliness questions from the social isolation battery will be used to measure loneliness with each question has a score ranging from 1 to 3 and a higher score indicates more loneliness.
Change in loneliness measured by a loneliness question. | Baseline to week 10
  The loneliness question will be used to measure perceived loneliness with a score ranging from 1 to 7 and a higher score indicates more loneliness.

SECONDARY OUTCOMES:
Change in attention | Baseline to week 10
  Attention is measured by using the Sustained Attention Response Task that involves pressing a button to frequently presented non-target trials (numbers 1, 2, 4, 5, 6, 7, 8, and 9) and withholding the button press to the infrequent target trials (number 3). The score (A prime) is calculated by considering accuracy on both non-target and target trials with a score maximum of 1. A higher score indicates better attentional performance.
Change in well-being as measured by the Perseverative Thought Questionnaire (PTQ) | Baseline to week 10
  PTQ is a 15-item questionnaire indexing the occurrence of negative thinking. The total PTQ score range is from 0 to 60, with a higher score indicating a frequent occurrence of negative thoughts.
Change in well-being as measured by the Experience of Intrusions Scale (EIS) | Baseline to week 10
  The EIS is a 5-item questionnaire indexing the impact of intrusive thoughts regarding an emotional event with a score ranging from 0 to 20. A higher score indicating a higher level of intrusions.
Change in well-being as measured by the short version of the perceived stress scale (PSS). | Baseline to week 10
  The short version of PSS is a 4-item questionnaire measuring the degree to which situations in one's life are viewed as stressful within the past month. The total score ranges from 0 to 16. A higher score indicates higher level of perceived stress.
Change in well-being as measured by the PERMA-Profiler | Baseline to week 10
  PERMA-Profiler a 15-item multidimensional measure used to index well-being according to the following 5 dimensions: positive emotions, engagement, relationships, meaning, and accomplishments. The score for each subscale range from 0 to 10, with a higher score indicating better well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Ninova, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No